CLINICAL TRIAL: NCT04216979
Title: Palmer's Point Versus The Umbilicus As Routine Primary Entry Site In Gynecologic Laparoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, basem mohamed hamed khalil, lecturer of obstetrics and gynecology/ MD ob/gyn, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5806-15-12-2019
Record Dates: First submitted 2019-12-19; First posted 2020-01-03 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-01

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- randomization (Experimental): Patients are randomly arranged in 2 groups Group (A):- Palmer's point is the primary entry site. Group (B):- The umbilicus is the primary entry site.
  Interventions: Procedure: laparoscopy entry policy
- group A (Experimental): these are the patient with palmars point as primary entry site
  Interventions: Procedure: laparoscopy entry policy
- group B (Experimental): these are the patient with umbilicus as primary entry site
  Interventions: Procedure: laparoscopy entry policy

INTERVENTIONS:
Procedure: laparoscopy entry policy — Patients will be randomly arranged in 2 groups Group (A):- Palmer's point is the primary entry site.
  Group (B):- The umbilicus is the primary entry site.

SUMMARY:
we will compare the classic method of using the umbilicus as the primary entry site in gynecological laparoscopy with Palmar's point

DETAILED DESCRIPTION:
All these cases will undergo:

1. History taking Patients are randomly arranged in 2 groups Group (A):- Palmer's point is the primary entry site. The stomach will be emptied of secretions and air following endotracheal intubation. (This is most easily performed using a nasogastric tube.) The left upper quadrant will be inspected for scars and the upper abdomen palpated for hepatomegaly or splenomegaly. A 10-mm incision will be made over Palmer's point. Veress needle first will be used for insufflation and tests of safety will be considered.

A 10-mm port will be held vertically and the layers observed via a 10-mm laparoscope. A gentle rotating action in a vertical direction was used to allow the bladeless tip to separate the tissues.

The layers of the abdominal wall seen at Palmer's point are as follows:

* skin,
* subcutaneous fat,
* external oblique aponeurosis,
* internal oblique aponeurosis,
* transversalis muscle fibres,
* (sometimes) extraperitoneal fat,
* peritoneum. Once the peritoneum will be breached, the introducer will be carefully removed from the port. The laparoscope will be then reintroduced.

An extra 360° check was then performed to exclude a through-and-through bowel injury. The umbilicus was then inspected and any adhesions cleared using one or more 5-mm ports inserted under direct vision. At the end of the operation, the skin was closed using a single subcuticular suture Group (B):- The umbilicus is the primary entry site. First of all, the umbilicus is well cleaned with a piece of gauze with betadine or alcohol then small incision is done (10mm) in the umbilicus, veress needle is then inserted and tests of safety of intraperotineal insufflation are considered. 10 mm port is then introduced with gentle rotating action in a vertical direction to allow the bladeless tip to separate the tissues.

The layers of the abdominal wall seen at Palmer's point are as follows:

* skin
* linea alba
* peritoneum. Once the peritoneum is breached, the trocar will be carefully removed from the port. The laparoscope will then reintroduced.

An extra 360° check was then performed to exclude a through-and-through bowel injury. At the end of the operation, the skin will be closed using a single subcuticular suture

ELIGIBILITY:
Inclusion Criteria:

* Patients listed for diagnostic or operative laparoscopy.

Exclusion Criteria:

* • Splenomegaly

  * Hepatomegaly
  * previous left upper quadrant surgery.
  * midline laparotomy
  * umbilical surgery
  * presence of umbilical hernia

Ages: 10 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Time assessed by the difference in using the umbilicus method as the primary entry site in gynecological laparoscopy with Palmar's point | 6 months
  the surgeon will calculate the time of surgery for similar cases in both groups and will compare between both groups according to the time factor
complications that occur in using the umbilicus method as the primary entry site in gynecological laparoscopy in comparison with Palmar's point | 6 months
  we will compare the number of participants with vascular or intestinal injuries in both procedures
coordination of the surgeon movement by the difference in using the umbilicus method as the primary entry site in gynecological laparoscopy in comparison with Palmar's point | 6 months
  questionnaire will be done to ask the surgeon about the degree of coordination and smoothness of using the surgeon his both hands in laparoscopy

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Zagazig University, Zagazig, East
  - Zagazig, Zagazig, East

IPD SHARING:
Plan to Share IPD: No